CLINICAL TRIAL: NCT00498719
Title: A Pilot Study of the Effectiveness of Cognitive Training in Preventing Attention Deficits Among Children in Treatment for Cancer
Brief Title: Cognitive Training in Attenuating Attention Deficits/Child Treatment for Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2004-0126
Record Dates: First submitted 2007-07-09; First posted 2007-07-10 (Estimated); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Leukemia; Lymphoma; Brain Tumor
Keywords: Leukemia; Lymphoma; Brain Tumor; Attention Deficit; Cognitive Training Program; Central Nervous System; CNS; CTP
MeSH Terms: conditions — Leukemia; Lymphoma; Brain Neoplasms; Attention Deficit Disorder with Hyperactivity | interventions — Cytidine Triphosphate; Control Groups

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CTP Group: One-on-one cognitive training
  Interventions: Behavioral: Cognitive Training Program
- Control Group: Standard educational support.
  Interventions: Other: Control Group

INTERVENTIONS:
Behavioral: Cognitive Training Program — Cognitive training sessions over a 4 to 6 month training period, each lasting about 2 hours.
  Other Names: CTP
  Groups: CTP Group
Other: Control Group — Standard educational support.
  Groups: Control Group

SUMMARY:
Primary Objectives:

1. To evaluate the feasibility of enrolling children and adolescents with newly diagnosed brain tumors, leukemia, or lymphoma in a program designed to prevent the academic and cognitive declines that commonly result following central nervous system (CNS) disease and treatment.

   Hypothesis 1: Despite the rigors of disease and treatment, children and adolescents will be able to participate in the CTP while they are receiving treatment for cancer. The high participation of our patients in routine school activities during treatment suggests that they will have the energy and interest required to participate in cognitive training.
2. To evaluate whether a Cognitive Training Program (CTP) might be helpful to patients in preventing attention deficits that commonly result following CNS disease and therapy.

   Hypothesis 2: Patients in the CTP arm of the study will show fewer declines in neurocognitive performance at the end of training and again six months later, as compared with the control group who will receive the usual services provided by the Education Program in Pediatrics.
3. To explore the relationship between CTP treatment compliance and stability/decline in cognitive and academic performance in children and adolescents who are being treated for brain tumors, leukemia, and lymphoma.

Hypothesis 3: Level of compliance with CTP treatment will be predictive of a patient's performance on neurocognitive measures.

DETAILED DESCRIPTION:
The Cognitive Training Program (CTP) is made up of many elements. It includes procedures that are designed to build five types of attention skills, as well as motivational activities that exercise your child's attention processes. The CTP includes instructions on how to improve the way your child's mind approaches a task, how he/she performs different tasks, and what he/she does after finishing tasks. The CTP also includes the use of therapy to improve and maintain motivation, self-esteem, and self-confidence, as well as to help your child stay motivated and keep from getting distracted.

Before your child can take part in this study, he/she will have what is called a "screening test of intelligence." This test will help the doctor decide if your child is eligible to take part in the study. In order for a child to participate in the study, he or she has to achieve a score > 70 on the screening test (at least within the borderline range of intelligence), because this level of intelligence is necessary for a child to understand the CPT educational materials. It is possible that after this test, your child may not be able to continue on this study. The screening test results will be discussed with you.

Your child will be randomly assigned (as in the toss of a coin) to either the CTP or a "control" group. The control group will receive standard educational support, but will not receive the one-on-one cognitive training given during the study. After the study is completed, patients randomized to the control group will be eligible to receive the CTP intervention, free of charge, if the parents prefer. All participants will complete standardized cognitive and academic tests at three time points: at the beginning of the study, six months later, and then six months after that. The tests will be given by a very experienced research assistant who will ask your child questions and have him or her complete various paper and pencil tasks or puzzles. Testing at each of the three time points will take about 3 hours. However, the test sessions can be divided into shorter sessions, if necessary for the child's comfort. After each test session, you and your child will talk to a member of the study staff about your child's results and what they mean to your child's progress.

Your child will be seen for a total of 20 study-therapy visits (as long as they are in the intervention group) over a 4 to 6 month training period. Each visit will be about two hours long, and will occur once a week during the training period. The study visits will be "one-on-one" sessions between your child and the therapist. Each study visit will be include two 50-minute training sessions with a 15-minute break between them. During training sessions, your child will participate in several activities. Each activity will only last about 15 minutes each. If your child gets tired during a session, the therapist will let him/her take a short rest break.

The therapy program your child receives will be especially designed for him/her, building on his/her strengths as well as focusing on areas where he/she needs more help.

This is an investigational study. CTP and assessment appointments will be scheduled on days that your child is already in the clinic or inpatient, as often as possible. About 30 children will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Eligibility criteria to participate in the study are: at least 6-years-old.
2. Enrolled in school or homebound instruction in a grade Kindergarten through 12th.
3. A diagnosis of leukemia, lymphoma, or brain tumor (e.g., primary brain tumors, leptomeningeal infiltration, or metastases) that requires treatment of the CNS (surgery, CRT, and/or chemotherapy).
4. Within 2 months to 14 months after beginning treatment for cancer.
5. Full scale IQ > or = 70.
6. English-speaking. (This is defined as the ability to appropriately respond to test and training materials.)

Exclusion Criteria:

1) A major physical, neurologic, or psychiatric condition that would preclude participation in the research program. The functional criteria for exclusion is inability to perceive and comprehend training materials and therapeutic interventions.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants with leukemia, lymphoma, or brain tumor that are at least 6 years old.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2004-04 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Academic + Cognitive Decline Pre- to Post-Treatment | 5 Years
  Determine whether Cognitive Training Program (CTP) prevents declines in cognitive and academic skills by comparing change from pre- to post-treatment through Academic achievement tests and psychological adjustment questionnaires at three points of time (baseline, at the end of training and 6 months later)

CONTACTS AND LOCATIONS:
Overall Officials: Martha Askins, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org